CLINICAL TRIAL: NCT05370053
Title: The Availability of the Enhanced Liver Fibrosis (ELF) Test Affects the Rate of Diagnosis of Nonalcoholic Steatohepatitis (NASH) With Fibrosis in Patients Referred to Hepatology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Winston Dunn, M.D., Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00145402
Record Dates: First submitted 2021-06-24; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Fatty Liver; NAFLD
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: During the hepatology evaluation for elevated liver enzymes or fatty liver at the University of Kansas Medical Center, the hepatologists (8 total) make a clinical decision on whether patients shall receive vibration-controlled transient elastography (VCTE). At the end of the clinic visit, patients were enrolled and randomized to receiving an enhanced liver fibrosis (ELF) test. If randomized to receiving the ELF testing, the hepatologist will receive the ELF result within 1 week. The hepatologist is free to the clinical information at hand to make clinical decisions. Possible decisions include: 1)defer liver biopsy without making a clinical diagnosis of cirrhosis 2)order liver biopsy, where the result may show F0-2 fibrosis, 3)order liver biopsy, where the result may show F3-4 fibrosis, 4)clinical diagnosis of cirrhosis without liver biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELF-test (Experimental): Patients receive ELF testing (a blood draw) and their hepatologist receives the result within a week.
  Interventions: Diagnostic Test: ELF Test
- Control (No Intervention): No intervention.

INTERVENTIONS:
Diagnostic Test: ELF Test — Patients receive ELF testing (a blood draw) and their hepatologist receives the result within a week.
  Arms: ELF-test

SUMMARY:
Background: During the hepatology evaluation, vibration-controlled transient elastography (VCTE) is often used as a clinical decision aid to target high-risk patients for liver biopsy. The enhanced liver fibrosis (ELF) test is expected to be approved in the US. We tested the hypothesis that making the ELF results available to the treating hepatologist will result in more appropriate and targeted use of liver biopsy in patients with elevated liver enzymes or fatty liver, and will result in more cases of advanced fibrosis/cirrhosis being diagnosed. Methods: During the hepatology evaluation for elevated liver enzymes or fatty liver at the University of Kansas Medical Center, the hepatologists (8 total) make a clinical decision on whether patients shall receive VCTE. At the end of the clinic visit, patients were enrolled and randomized to receiving an ELF test. Patients with liver biopsy within the last five years or decompensated cirrhosis were excluded. The primary outcome is the rate of a diagnosis of F3-4 fibrosis based on liver biopsy or clinical diagnosis of cirrhosis with the initiation of hepatocellular carcinoma surveillance. Four hundred fifty patients are to be enrolled over two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients from hepatology clinic undergoing new evaluation for NAFLD.

Exclusion Criteria:

* Patients with liver biopsy within the last five years or decompensated cirrhosis were excluded. Patients known to have other liver diseases were also excluded. Patients consuming > 14 drinks in the past 6 months were excluded. Patients may be subsequently found to have positive viral or autoimmune serologies after enrollment because the serology result is typically not available at the time of enrollment. These patients will be excluded from the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
A diagnosis of F3-4 fibrosis based on liver biopsy or clinical diagnosis of cirrhosis. | 2 years
  The number of patients diagnosed with stage 3-4 based on liver biopsy or clinical diagnosis of cirrhosis in each arm of the study.
  Clinical diagnosis of cirrhosis is defined as provider diagnosing cirrhosis and ordering of hepatocellular carcinoma surveillance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States